CLINICAL TRIAL: NCT05690971
Title: Randomized Controlled Trial of a Psychosocial Mobile Application (App) to Promote Coping for Patients With Chronic Graft-Versus-Host Disease (GVHD)
Brief Title: Psychosocial Mobile App for Chronic Graft-Versus-Host Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-503
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Graft-Versus-Host Disease; Allogeneic Stem Cell Transplant
Keywords: Chronic Graft-Versus-Host Disease; Allogeneic Stem Cell Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Horizons mobile app (Experimental): Participants randomly assigned to the Horizons group, will use the Horizons app over an eight-week period in addition to receiving usual care from transplant team.
  Participants will complete study questionnaires at the time of enrollment (baseline) and at eight and sixteen weeks after enrollment
  Interventions: Behavioral: App
- Usual Care (Active Comparator): Participant in the usual care group will receive usual care from the transplant oncology team including all the supportive care measures implemented by the transplant oncology team.
  Participants will complete study questionnaires at the time of enrollment (baseline) nad at eight and sixteen weeks after enrollment
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: App — HORIZONS is self-administered with several features to promote engagement and health behavior change including gamification strategies, videos of chronic GVHD survivors, and optional content.
  HORIZONS includes five interactive modules to be completed during an eight week period. HORIZONS also includes a sixth optional helpful resources section with a review of the domains and skills covered in the first five modules
  Arms: Horizons mobile app
Behavioral: Usual Care — Patients in the usual care group will receive usual care from the transplant oncology team including all the supportive care measures implemented by the transplant oncology team.
  Arms: Usual Care

SUMMARY:
The purpose of this research study is to see whether a psychosocial mobile app called Horizons is effective at improving quality of life, symptom burden, psychological distress, and coping in patients living with chronic graft-versus host disease (GVHD)

DETAILED DESCRIPTION:
Frequently patients living with chronic GVHD experience physical and emotional symptoms during the course of illness that impacts their quality of life. Patients also often report difficulty managing many of the tasks they need to do to manage their chronic GVHD. They also frequently have a lot of questions about chronic GVHD and the expected trajectory of this illness.

The purpose of this research study is to see whether a psychosocial mobile app called Horizons is effective at improving quality of life, symptom burden, and psychological distress in patients with chronic GVHD

* This study will randomly assign participants to either receiving Horizons plus usual care or usual care alone.
* Enrolled participants will be on the research study for up to sixteen weeks and it is expected that about 120 people will take part in this research study.

The Leukemia and Lymphoma Society is supporting this research by providing funding.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who underwent allogeneic hematopoietic stem cell transplant (HCT).
* Have moderate to severe chronic GVHD based on their oncology clinician assessment as documented in the Electronic Health Record.
* Ability to comprehend and speak English as the HORIZONs app is only available in English.

Exclusion Criteria:

-Patients with acute or unstable psychiatric or cognitive conditions which the treating clinicians believes prohibits informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QOL): Functional Assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) | 8 Weeks
  Compare patient QOL (FACT-BMT) between usual care and Horizon at 8 weeks using ANCOVA. FACT-BMT score range 0-164, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Quality of life (QOL) longitudinal using FACT-BMT | Up to sixteen weeks
  Compare patient QOL (FACT-BMT) longitudinally between Horizons and usual care group using mixed linear effect models. FACT-BMT score range 0-164, with higher scores indicating better quality of life.
Anxiety symptoms using the Hospital Anxiety and Depression Scale (HADS-Anxiety) | up to sixteen weeks
  Compare anxiety symptoms (HADS-Anxiety) between study groups. The HADS anxiety subscale range from 0-21 with higher scores indicating worse anxiety symptoms
Depression symptoms using HADS-Depression | up to sixteen weeks
  Compare depression symptoms (HADS-depression) between study groups. The HADS depression subscale range from 0-21 with higher scores indicating worse depression symptoms
Chronic GVHD symptom burden (Lee Scale) | up to sixteen weeks
  compare chronic GVHD symptom burden (Lee Scale) between the study groups. The Lee Scale ranges from 0-100 with higher scores indicating worse symptom burden

OTHER OUTCOMES:
Self-efficacy (PROMIS self-efficacy scale) | up to sixteen weeks
  Compare self-efficacy (PROMIS-self-efficacy scale) between the study groups. The PROMIS self-efficacy for managing symptoms scale ranges from 0-100 with higher scores indicating better self-efficacy
patient coping using Measure of Current Status (MOCS) | up to sixteen weeks
  Comparing coping (MOCS) between study groups (MOCS score range 0-52, with higher scores indicating greater coping skill).
social support using Medical Outcomes Study Social Support Survey (MOS SSS) | up to sixteen weeks
  Compare patient social support (MOS SSS) between study groups. MOS SSS score range 0-100, with higher scores indicating greater support.
Usability of the Horizons app using the system usability scale | eight weeks
  We will use the system usability scale at 8 weeks post-intervention (for those randomized to Horizons) to assess the usability of HORIZONS. the system usability scale score range from 0-100 with higher scores indicating better usability

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation